CLINICAL TRIAL: NCT03833232
Title: Omentopexy With Glubran®2 for Reducing Complications After Laparoscopic Sleeve Gastrectomy: Results of a Prospective Study.
Brief Title: Omentopexy With Glubran®2 for Reducing Complications After Sleeve Gastrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Salerno (Other)
Responsible Party: Principal Investigator, SALVATORE TRAMONTANO, Clinical Professor, University of Salerno
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110511
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Obesity With BMI >35

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omentopexy and cyanoacrilate glue (Experimental): Apposition of omentum with cyanoacrilate glue after gastric section
  Interventions: Device: omentopexy with cyanoacrilate glue
- gastrectomy without omentopexy (No Intervention): Gastric section without omentopexy

INTERVENTIONS:
Device: omentopexy with cyanoacrilate glue — apposition of omentum with cyanoacrilate glue on gastric section
  Other Names: omentopexy with Glubran 2
  Arms: omentopexy and cyanoacrilate glue

SUMMARY:
BACKGROUND. Gastric fistulas, bleeding, and strictures are commonly reported after laparoscopic sleeve gastrectomy (LSG), that increase morbidity and hospital stay and may put the patient's life at risk. This trial reports our prospective evaluation of application of synthetic sealant, a modified cyanoacrylate (Glubran®2), on suture rime, associated with omentopexy, to identify results on LSG-related complications.

METHODS. Patients were enrolled for LSG by two Bariatric Centers, with high-level activity volume. Intraoperative recorded parameters were: operative time, estimated intraoperative bleeding, conversion rate. Presence of early complications after LSG during the follow up period was evaluated. Overall complications were analyzed. Perioperative data and weight loss were also evaluated. A control group was identified for the study.

DETAILED DESCRIPTION:
The prospective randomized trial is designed with the aim to verify the effectiveness of the Glubran®2 used in its spray application, according to manufacturer's indications, to perform the omentopexy of the staple line to prevent and reduce early complications after LSG. single-blind randomization was explained: a single surgeon, in enrollment phase, assigned patient to case or control group, after adequate communication of randomization to all patients. The surgeon that performed procedure only knew if patient was randomized to case group (LSG with omentopexy with Glubran®2) or to control group (LSG without omentopexy with Glubran®2). Control group was identified for the study with simple randomization, considering patients treated with LSG during same period. Patients of case and control groups were not paired. Same recording was performed for both groups. Patients were enrolled for LSG by two Bariatric Centers, with high-level activity volume, after multidisciplinary evaluation: inclusion criteria, according with international guidelines, was body mass index (BMI) of greater than 40 kg/m2 or > 35 with at least one co-morbidity, such as hypertension, dyslipidemia or diabetes, age ≥ 18 years old, medically unfit for surgical intervention, absence of active gastric disease, of uncontrolled medical or psychiatric conditions, and signed informed consent. Bariatric procedure was performed according with standardized four-trocars technique. All surgeons involved had a proved experience for bariatric surgery, and have completed learning curve.

The size of the boogie to be used for calibration ranged from 42 to 48 Fr, among two groups. In case group, after gastric partition and confirming correct closure of mechanical section (performed with Endo-Gia, varying depth of stapler, from 3.5 mm blue to 4.4 black charge, according with gastric level), a layer of the synthetic sealant on all rime suture was applied and an omentum flap to place was apposed. Absence of gastric rotation with omentum flap, or any tension on the resected stomach was carefully controlled. In control group, we reinforced staple line with buttressing (bovine pericardium) of mechanical stapler, or with running suture of the rime alone, indifferently. A recording of type of reinforcing was performed, also if not pertinent to study.

Anthropometric data recorded were: age, weight, BMI, presence of comorbidities. Intraoperative recorded parameters were: operative time, estimated intraoperative bleeding (in ml), conversion rate. We prospectively evaluated the presence of early complications after LSG during the follow up period (30 days from intervention). Considered complications were staple line leakage/gastric fistula, postoperative bleeding, intraabdominal abscess, cardiopulmonary failure, and all other complications. In order to considering effects and real impact of mentioned events, we also evaluated length of hospital stay, rate of readmission, rate of reintervention, overall mortality at 30 days. Weight loss was recorded at 15 and 30 days, as excess weight loss percent (EWL%) and as reduction of BMI.

The demographic data and perioperative data were compared using the student's t and Mann- Whitney U tests for continuous variables. Fisher's exact test was used to determine any statistical significance for the categorical variables. The continuous variables were presented as mean ± standard deviation and the categorical variables were presented as the number (%). The level of significance was set at 0.05.

All procedures involving human participants were in accordance with the Ethical standards of the institutional research committee and with the 1964 Helsinki declaration and its later amendments.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) of greater than 40 kg/m2 or > 35 with at least one co-morbidity, such as hypertension, dyslipidemia or diabetes,
* age ≥ 18 years old,
* medically unfit for surgical
* absence of active gastric disease, of uncontrolled medical or psychiatric conditions,
* signed informed consent.

Exlusion criteria

- patient not suitable for bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
fistulization rate | 12 months

SECONDARY OUTCOMES:
bleeding rate | 12 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pilone V, Tramontano S, Renzulli M, Romano M, Monda A, Albanese A, Foletto M. Omentopexy with Glubran(R)2 for reducing complications after laparoscopic sleeve gastrectomy: results of a randomized controlled study. BMC Surg. 2019 Nov 5;19(Suppl 1):56. doi: 10.1186/s12893-019-0507-7. PMID 31690312